CLINICAL TRIAL: NCT01221636
Title: A Study to Compare the Pharmacokinetics of Abatacept (BMS-188667) Drug Product Using Active Pharmaceutical Ingredient Manufactured With a High Concentration of Metals Relative to the Active Pharmaceutical Ingredient Manufactured With a Low Concentration of Metals
Brief Title: Pharmacokinetic Study to Compare the Blood Levels of Low vs High Metal Manufacture of Abatacept
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IM101-278
Record Dates: First submitted 2010-10-13; First posted 2010-10-15 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2011-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Metal Abatacept (Other): Reference
  Interventions: Drug: Abatacept
- High Metal Abatacept (Experimental)
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — Solution for injection, Intravenous, 750 mg, 1 day
  Other Names: Orencia; BMS-188667

SUMMARY:
The purpose of this study is to determine whether the blood levels of abatacept drug product manufactured using High Metals and using Low Metals are comparable in healthy subjects.

DETAILED DESCRIPTION:
Compare the pharmacokinetic (PK) of High Metals abatacept relative to Low Metals abatacept following a single intravenous infusion of 750 mg in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations
* Body weight will be between 60 and 100 kg, inclusive

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Any major surgery within 4 weeks of study drug administration
* Smoking more than 10 cigarettes per day
* Recent (within 6 months of study drug administration) drug or alcohol abuse
* Positive blood screen for hepatitis C antibody, hepatitis B surface antigen, or HIV-1, -2 antibody
* History of any significant drug allergy or asthma
* Women who are pregnant or breastfeeding and/or unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Single-dose pharmacokinetic parameters: Cmax (Maximum observed serum concentration) | Over 71 days after single dose administered
Single-dose pharmacokinetic parameters: AUC 0-71 days (Area under the serum concentration-time curve from time zero to 71 days) | Over 71 days after single dose administered
Single-dose pharmacokinetic parameters: AUC (INF) (Area under the serum concentration-time curve from time zero extrapolated to infinity) | Over 71 days after single dose administered

SECONDARY OUTCOMES:
Immunogenicity determination will be based on titers of anti abatacept and anti-CTLA-4-T antibodies in serum over time | Days 29, 57, and 71 after single dose administered
Safety assessments: adverse events, vital sign measurements, ECGs, physical examinations, and clinical laboratory tests. The incidence of observed adverse events will be tabulated and reviewed for potential significance and clinical importance | Days 1, 2, 4, 8, 15, 22, 29, 43, 57 and 71 after single dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Austin, Texas, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx